CLINICAL TRIAL: NCT07230132
Title: A Multicenter, Randomized, Double-blind, Placebo-controlled Study to Evaluate the Efficacy and Safety of Various Doses of ZT006 in Overweight and Obese Participants
Brief Title: Efficacy and Safety of ZT006 in Overweight and Obese Participants
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Beijing QL Biopharmaceutical Co.,Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BJQL-ZT006-2001
Record Dates: First submitted 2025-11-13; First posted 2025-11-17 (Actual); Last update posted 2025-11-17 (Actual); Status verified 2025-09

CONDITIONS: Overweight , Obesity
MeSH Terms: conditions — Overweight; Obesity

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- ZT006 tablet low target dose (Experimental): administered per os, daily
  Interventions: Drug: ZT006
- ZT006 tablet medium target dose (Experimental): administered per os, daily
  Interventions: Drug: ZT006
- ZT006 tablet high target dose (Experimental): administered per os, daily
  Interventions: Drug: ZT006
- placebo of ZT006 (Placebo Comparator): administered per os, daily
  Interventions: Drug: Placebo of ZT006

INTERVENTIONS:
Drug: ZT006 — Participants will receive a daily dose of ZT006
  Arms: ZT006 tablet high target dose; ZT006 tablet low target dose; ZT006 tablet medium target dose
Drug: Placebo of ZT006 — Participants will receive a daily dose of placebo of ZT006
  Arms: placebo of ZT006

SUMMARY:
This study is being conducted to evaluate the efficacy and safety of ZT006 tablet in participants with overweight and obesity.

In addition to dietary caloric restriction and increased physical activity, study participants will receive either ZT006 tablets or placebo tablets once every morning (placebo looks like ZT006 tablets but has no active pharmaceutical ingredients). For a fair comparison, study participants are assigned to ZT006 or placebo randomly by a computer.

The treatment will last for 28 weeks. ZT006 tablets will be administered in an up-titration fashion, i.e. the dose of ZT006 will be gradually increased to reach three target doses so that the participants can tolerate its effect. Participants will have 17 clinic visits including one screening visit and one follow-up visit.

Female participants who are pregnant, breast-feeding or who plan to become pregnant during the study are not allowed to participate in the study. Pregnancy will be checked by blood or urine tests during the study.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, age between 18 - 65 years (both inclusive) at the time of signing of the informed consent.
* Body mass index (BMI) greater than or equal to 28 kg/m², or greater than or equal to 24 kg/m²with at least one of the comorbidities: hypertension, hyperlipidemia, pre-diabetes, metabolic dysfunction-associated steatotic liver disease (MASLD) or obstructive sleep apnea-hypopnea syndrome (OSAHS).
* Having dietary caloric restriction and increased physical activity for ≥3 months, with change in body weight (increase or decrease) no more than 5%, irrespective of medical records.

Exclusion Criteria:

* Type 1 or type 2 diabetes or other specific types derived from other causes
* Medical history of acute or chronic pancreatitis
* Medical history of cholecystitis, gallstone ≤1 cm, or history of symptomatic gallbladder diseases
* Use of glucagon-like peptide-1 (GLP-1) agonist, dual GLP-1/glucose-dependent insulinotropic polypeptide (GIP) or GLP-1/glucagon agonist, or triple GLP-1/GIP/glucagon agonist within 90 days before screening
* HbA1c ≥ 6.5% or fasting plasma glucose ≥ 7.0 mmol/L at screening
* Triglyceride ≥ 5.7 mmol/L at screening
* Calcitonin ≥ 50 ng/L at screening

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2025-12 (Estimated); Primary Completion 2026-12 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
Change in body weight relative to baseline | Percentage-point from baseline to end of treatment (week 28)
  Percentage-point

SECONDARY OUTCOMES:
Proportion of participants who achieved body weight reduction greater than or equal to 5% at week 28 | From baseline to end of treatment (week 28)
  Proportion of participants in %
Proportion of participants who achieved body weight reduction greater than or equal to 10% at week 28 | From baseline to end of treatment (week 28)
  Proportion of participants in %
Proportion of participants who achieved body weight reduction greater than or equal to 15% at week 28 | From baseline to end of treatment (week 28)
  Proportion of participants in %
Change in body weight | From baseline to end of treatment (week 28)
  Measured in kg
Change in waist circumference | From baseline to end of treatment (week 28)
  Measured in cm
Change in body mass index (BMI) | From baseline to end of treatment (week 28)
  Measured in kg/m²（ Body weight in kilogram divided by the square of height in meter ）
Rate of treatment-emergent adverse events | From baseline to end of study (week 33)
  Summarized from adverse event reporting in %
Rate of serious adverse events | From baseline to end of study (week 33)
  Summarized from adverse event reporting in %
Proportion of participants with positive anti-ZT006 antibody | From baseline to end of treatment (week 33)
  Summarized in %

CONTACTS AND LOCATIONS:
Overall Officials: Linong Ji, MD, Principal Investigator — Peking University People's Hospital
Locations (10):
- China (10):
  - Handan First Hospital, Handan, Hebei
  - Hebei Petro China Cental Hospital, Langfang, Hebei
  - Harbin Medical University Affiliated Fourth Hospital, Harbin, Heilongjiang
  - Luoyang Third People's Hospital, Luoyang, Henan
  - YueYang People's Hospital, Yueyang, Hunan
  - The Second Affiliated Hospital of Nanjing Medical University, Nanjing, Jiangsu
  - Central Hospital Affiliated to Shandong First Medical University, Jinan, Shandong
  - First Hospital of Shanxi Medical University, Taiyuan, Shanxi
  - Xi'an Daxing Hospital, Xi’an, Shanxi
  - Peking University People's Hospital, Beijing